CLINICAL TRIAL: NCT00228306
Title: Effect of Cardiovascular Fitness on Motor Learning and Executive Function in Individuals After Stroke
Brief Title: The Effect of Aerobic Exercise on Learning After Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9903; Am Heart Assn 0530208N
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Rehabilitation exercise
- 2 (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Rehabilitation exercise — Rehab therapy is delivered for 8 weeks.
  Arms: 1

SUMMARY:
Determine if attaining aerobic fitness is beneficial in producing cortical neuroplasticity in individuals with chronic stroke.

DETAILED DESCRIPTION:
Crossover clinical trial. Experimental group undergoes 3x/wk/6 months of aerobic conditioning. Control group performs usual daily activities. All participants will be assessed with cognitive and motor behavioral testing at baseline, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Single ischemic stroke occuring 6-72 months prior
* Fugl-Meyer score (upper + lower extremity) 45 or greater
* Mini mental status score of >23
* approval of the subject's medical doctor

Exclusion Criteria:

* already performing >20 min of cardiovascular exercise 3x/wk or more
* alcohol consumption of >2 oz. liquor, 8 oz. wine or 24 oz beer/day
* cardiac history of unstable angina, recent myocardia infarction within the last 3 months, congestive heart failure, significant valve dysfunction
* medical history of recent hospitalization (> 3 months) for medical illness
* symptomatic peripheral arterial occlusive disease
* orthopedic or chronic pain conditions restricting exercise
* pulmonary or renal failure
* active cancer
* unstable hypertension (>160/100 mmHg)
* diabetes mellitus (fasting glucose > 180 NG./dk, HgA1C > 10%) that is unable to be controlled < month
* receptive or expressive aphasia as indicated on MMSE
* multiple strokes or other neuromuscular conditions
* major depression that is untreated using the Beck depression inventory

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Motor learning behavioral measures; executive function behavioral measures. | Baseline, 8 weeks, 12 weeks

SECONDARY OUTCOMES:
Peak V02 and other aerobic capacity measures. Physical disability measures. | Baseline, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Quaney, PT, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States